CLINICAL TRIAL: NCT02501733
Title: Medacta GMK Sphere® Medial Pivot, Cruciate Substituting Multicenter, Post-Market Outcomes Study
Brief Title: Medacta GMK Sphere® Multicenter Post-Market Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121416-01
Record Dates: First submitted 2015-06-25; First posted 2015-07-17 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
Keywords: Total Knee Replacement; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medacta GMK Sphere® Knee Prosthesis (Other): All subjects enrolled will receive the Medacta GMK Sphere® Medial Knee Prosthesis
  Interventions: Device: Medacta GMK Sphere® Medial Knee Prosthesis

INTERVENTIONS:
Device: Medacta GMK Sphere® Medial Knee Prosthesis — There is no consensus within the Arthroplasty community as to whether a traditional post and cam-style Posterior Stabilized total knee device is superior to a medial-pivot, more congruent device. However, the majority of surgeons seem to prefer the former, though there is a minority that uses the latter device with great success.
  To date, there have been few prospective trials directly comparing these devices, and none with the latest generation of Total Knee Arthroplasty implants. Almost all such studies have been retrospective and/or utilizing older generation devices.
  Other Names: Total Knee Arthroplasty; Total Knee Prosthesis

SUMMARY:
This study is to average Forgotten Knee Score (FJS) of those patients receiving the Medacta GMK Sphere® knee at the two and five year time points. 70 subjects, enrolled at the data coordinating center in Medacta GMK Sphere® vs Posterior Stabilized study (WIRB Pro Num: 20141994) and randomized to the Sphere arm, will have their data utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the informed consent
* Patients able to comply with follow-up requirements including postoperative weight bearing restrictions and self evaluations.
* Male and non-pregnant female patients ages 21 - 80 years of age at the time of surgery.
* Patients requiring a primary total knee replacement.
* Patients with a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
* Patients with intact collateral ligaments.

Exclusion Criteria:

* Patients with inflammatory arthritis.
* Patients that are morbidly obese, body mass index (BMI) > 40.
* Patients with a history of total or unicompartmental reconstruction of the affected joint.
* Patients that have had a high tibial osteotomy or femoral osteotomy.
* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
* Patients that are immunologically compromised, or receiving chronic steroids (> 30 days).
* Patients bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
* Patients with knee fusion to the affected joint.
* Patients with an active or suspected latent infection in or about the knee joint.
* Patients that are prisoners.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in Forgotten Knee Scores (FJS) of those patients receiving the Medacta GMK Sphere from baseline to years 2 and 5 post-operatively. | Baseline, 2 and 5 year time points
  Knee function-patients ability to forget the artificial joint in everyday life.

SECONDARY OUTCOMES:
Total Knee Society Score (KSS) | Pre-operative, 6 weeks, 3-6 months, 1,2,3,4 and 5 years.
  Total Knee Society score questionnaire to assess pain and function
Krackow Activity Scale (KAS) | Pre-operative, 6 weeks, 3-6 months, 1,2,3,4 and 5 years
  The Krackow Activity Scale (KAS) lower extremity activity scale.
Radiographic Analysis | Pre-operative, 6 weeks, 3-6 months, 1,2,3,4 and 5 years
AP long standing X-ray | Pre-operative and 6 weeks
  Determine degree of Varus or Valgus

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Norhtwestern University, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - McBride Orthopedic Hospital, Oklahoma City, Oklahoma
  - Texas Orthopedics, Austin, Texas
  - Spokane Joint Replacement Center, Spokane, Washington